CLINICAL TRIAL: NCT00633789
Title: A Randomized Discontinuation Study of Brivanib Alaninate (BMS-582664) Versus Placebo in Subjects With Advanced Tumors
Brief Title: Phase II Study of Brivanib (BMS-582664) to Treat Multiple Tumor Types
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CA182-026
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Advanced Non-small Cell Lung Cancer; Transitional Cell Carcinoma; Soft Tissue Sarcoma; Gastric/Esophageal Adenocarcinoma; Pancreatic Cancer Including Ampulla of Vater
MeSH Terms: conditions — Carcinoma, Transitional Cell; Sarcoma; Adenocarcinoma Of Esophagus | interventions — brivanib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: brivanib
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: brivanib — Tablets, Oral, 800 mg, once daily, until progression
  Other Names: BMS-582664
  Arms: 1
Drug: Placebo — Tablets, Oral, 0 mg, once daily, until progression
  Arms: 2

SUMMARY:
The purpose of this study is to determine if gastric/esophageal, lung, pancreatic, bladder and sarcoma patients show benefit from brivanib treatment. Patients who clearly do, stay on treatment. Those in which it is unclear will be randomized to continue or withdraw treatment to determine whether that benefit is related to brivanib

ELIGIBILITY:
For additional information, please contact the BMS oncology clinical trial information service at 855-216-0126 or email MyCancerStudyConnect@emergingmed.com. Please visit www.BMSStudyConnect.com for more information on clinical trial participation.

Inclusion Criteria:

* Life expectancy at least 3 months
* Diagnosis of a solid tumor which is unresectable in which no approved effective therapy exists or for subjects who are intolerable to such therapy. The initial enrollment will focus on non-small cell lung, gastric/esophageal adenocarcinoma, soft tissue sarcoma, transitional cell carcinoma, and pancreatic cancer including ampulla of Vater tumors
* Adequate tumor sample
* Adequate recovery (baseline or Grade 1) from recent therapy. At least 1 week must have elapsed from the time of a minor surgery, and at least 8 weeks for major surgery or radiation therapy

Exclusion Criteria:

* Subjects with known brain metastasis.
* Subjects with signs or symptoms suggestive of brain metastasis are not eligible unless brain metastases are ruled out by CT or MRI

Medical History and Concurrent Diseases:

* History of thrombo-embolic disease within the last six months requiring therapeutic anticoagulation
* Subjects with history of poor wound healing or non healing ulcers
* Uncontrolled or significant cardiovascular disease

Allergies and Adverse Drug Reactions:

* History of allergy to brivanib its drug class, or related compounds

Prohibited Treatments and/or Therapies:

* Exposure to any investigational drug within 4 weeks of enrollment
* Other concurrent chemotherapy, hormonal therapy, immunotherapy regimens or radiotherapy, standard or investigational. Subjects may continue to receive hormone replacement therapy
* Prior exposure to brivanib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 597 (Actual)
Dates: Start 2008-06; Primary Completion 2012-02 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Radiographic imaging and clinical evaluation will be used for tumor assessment | every 6 weeks

SECONDARY OUTCOMES:
Safety profiles | ongoing throughout trial
Disease response rate | determined June 2010
Disease control rate | determined June 2010
Pharmacokinetics | determined June 2010
Pharmacodynamics | determined June 2010
Biomarkers | determined June 2010

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (20):
- United States (6):
  - University Of Chicago, Chicago, Illinois
  - Northshore Univ. Healthsystem, Evanston, Illinois
  - Sidney Kimmel Comprehensive Cancer Center At Johns Hopkins, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Ctr, New York, New York
  - University Of Pennsylvania, Philadelphia, Pennsylvania
- Argentina (2):
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
- Local Institution, Brussels, Belgium
- Canada (2):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Toronto, Ontario
- Local Institution, Paris, France
- Germany (2):
  - Local Institution, Freiburg im Breisgau
  - Local Institution, Halle
- Netherlands (3):
  - Local Institution, Maastricht
  - Local Institution, Rotterdam
  - Local Institution, Utrecht
- Local Institution, Gdansk, Poland
- United Kingdom (2):
  - Local Institution, Glasgow, Scotland, Strathclyde
  - Local Institution, Surrey

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx